CLINICAL TRIAL: NCT05656846
Title: The Effect of Biweekly Follow up Along With at Home Ultrasound on the Anxiety of Pregnant Women Following Recurrent Pregnancy Loss.
Brief Title: Biweekly Follow-Up and At-Home Ultrasound Reduce Anxiety in Women With Recurrent Pregnancy Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Michal Levy, MD, Principal Investigator, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: WOMC-0130-22
Record Dates: First submitted 2022-10-20; First posted 2022-12-19 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Recurrent Pregnancy Loss

STUDY DESIGN:
Intervention Model Description: 1. Recruitment of eligible patients. Patients will receive an explanation of the study protocol, purpose and methodology including the difference between the two study groups. Willing participants will sign an informed consent.
  2. Initiation visit, the patient will be randomly assigned to one of the 2 study groups.
  3. Following the random assignment, all participants will complete 3 validated questionnaires.
     Addendum 1. Questionnaire: Maternal Antenatal Attachment Scale-MAAS (female) Addendum 2. Revised Prenatal Distress Questionnaire. Addendum 3. After completion of the questionnaires, patients will be instructed on the mode of operation of home ultrasound device (pulsenmore), the frequency and means of communication with the study team.
  4. At 20-22 weeks of gestation, completion of the three questionnaires.
  5. Collected data
     1. Demographic characteristics
     2. Antenatal follow-up
     3. Results of the various questionnaires
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: PulseNmore ES™ (Experimental): Experimental: PulseNmore ES™:
  The study population will be recruited between 12 and 14 weeks of gestation. These patients will be followed using a twice weekly virtual visit by a member of the study team. This visit will include a short survey of obstetrical complaints such as contractions leakage of fluid and decreased fetal movements, as well as a brief sonographic survey using the portable ultrasound device.
  Interventions: Device: PulseNmore ES™
- Control Standard Ultrasound (Active Comparator): A population of patients between 12 and 22 weeks of gestation with history of recurrent pregnancy losses who will be subjected to routine antenatal care as per clinic protocol. These patients will not receive the additional intervention.
  Interventions: Device: Standard Ultrasound

INTERVENTIONS:
Device: PulseNmore ES™ — The patients will be instructed on the mode of operation of home ultrasound device (pulsenmore), the frequency and means of communication with the study team.
  Arms: Experimental: PulseNmore ES™
Device: Standard Ultrasound — These patients will not receive the additional intervention and will use the Standard Ultrasound. A population of patients between 12 and 22 weeks of gestation with history of recurrent pregnancy losses who will be subjected to routine antenatal care as per clinic protocol. These patients will not receive the additional intervention.
  Arms: Control Standard Ultrasound

SUMMARY:
Spontaneous pregnancy loss is a relatively common phenomenon, with 10-15% of clinically recognized pregnancies ending in miscarriage.1 Recurrent pregnancy loss (RPL) is a disorder defined by two or more failed pregnancies2. According to various studies, pregnancy loss has been described as a traumatic event for couples even if the loss occurs at a very early stage of pregnancy.

Few controlled studies dealt with the effects of the miscarriage on the psychological condition of women during a subsequent pregnancy, 4,6-8.

This study aimed to evaluate the effectiveness of "at home ultrasound" in addition to routine prenatal care in reducing maternal anxiety during pregnancy for patients with history of recurrent pregnancy loss.

i. Inclusion criteria:

1. Patients with recurrent pregnancy losses in first trimester
2. Current pregnancy gestational age 12-14 week of gestation
3. Singleton pregnancy ii. Exclusion criteria:

1. Female subjects who refuse to participate 2. Female subjects who don't speak Hebrew

Device details:

Pulsenmore Specifications:

Compatible with: Android mobile phones with USB type C connector (Samsung S8+, Nokia 8, Nokia 7.1) ApplicatThe aim of this study is to evaluate the effectiveness of "at home ultrasound" in addition to routine prenatal care in reducing maternal anxiety during pregnancy for patients with history of recurrent pregnancy loss.ion: PulseNmore ES™, downloadable from Google Play™ Store.

DETAILED DESCRIPTION:
Background:

Spontaneous pregnancy loss is a relatively common phenomenon, with 10-15% of clinically recognized pregnancies ending in miscarriage.1 Recurrent pregnancy loss (RPL) is a disorder defined by two or more failed pregnancies2. According to various studies, pregnancy loss has been described as a traumatic event for couples even if the loss occurs at a very early stage of pregnancy.3-5 Few controlled studies dealt with the effects of the miscarriage on the psychological condition of women during a subsequent pregnancy4,6-8. These studies establish proof of considerably increased pregnancy specific anxiety in pregnant women with a history of spontaneous abortion, compared to pregnant women with no history of spontaneous abortion. As in the study of Bergner et al. women after early miscarriages are under pressure in a new pregnancy due to emotional disorders in the shape of pregnancy-specific anxiety, mostly before the critical point in the pregnancy when the previous miscarriage took place is passed.6 In order to offer pregnant women who have previously suffered miscarriages, apart from adequate psychological support alongside workup to find the RPL etiology, some reassurance and comfort this study aimed to evaluate the effectiveness of "at home ultrasound" in addition to routine prenatal care in reducing maternal anxiety during pregnancy for patients with history of recurrent pregnancy loss.

Study primary objectives/hypotheses:

Of all interventions that can alleviate the stress during pregnancy, we wish to learn the effect of "at home ultrasound" used by patients and feedback by clinician.

The aim of this study is to evaluate the effectiveness of "at home ultrasound" in addition to routine prenatal care in reducing maternal anxiety during pregnancy for patients with history of recurrent pregnancy loss. We hypothesize that couples would feel calmer and more reassured regarding their pregnancy.

Administrative Organization:

Department of Obstetrics and Gynecology at the Edith Wolfson Medical Center, Holon, Israel.

Study population The study population includes gravid patients recruited between 12 weeks of gestation and 14 weeks. Eligible patients include women with recurrent pregnancy losses in first trimester. This is a randomized controlled prospective trial registered at TRIALS.GOV The study population will be recruited between 12 and 14 weeks of gestation. The study population will be subject to standard routine antenatal care per clinic protocol. In addition, these patients will be followed using a twice weekly virtual visit by a member of the study team. This visit will include a short survey of obstetrical complaints such as abdominal pain and vaginal bleeding, as well as a brief sonographic survey using the portable ultrasound device. The details and findings of the visit will be recorded in the medical charts. The portable device will be handed to the patient during the intake visit of the study. The patient will be instructed how to operate the device by a team member.

Pulsenmore Specifications:

Compatible with: Android mobile phones with USB type C connector (Samsung S8+, Nokia 8, Nokia 7.1) Application: PulseNmore ES™, downloadable from Google Play™ Store

Network Connectivity: Wi-Fi or cellular (via user's mobile phone) Data Upload: Secured cloud service compliant with formal information security standards and directives Probes used only for external use on intact skin without contamination of blood or bodily fluids and should be cleaned with low-level disinfection between each use and sterilized prior patient exchange according to our departmental protocol.

The control group: A population of patients between 12 and 22 weeks of gestation with history of recurrent pregnancy losses who will be subjected to routine antenatal care as per clinic protocol. These patients will not receive the additional intervention.

i. Inclusion criteria:

1. Patients with recurrent pregnancy losses in first trimester
2. Current pregnancy gestational age 12-14 week of gestation
3. Singleton pregnancy ii. Exclusion criteria:

1. Female subjects who refuse to participate 2. Female subjects who don't speak Hebrew

Methods:

1. Recruitment of eligible patients will be conducted during routine visits to the maternal fetal outpatient clinic. Patients will receive an explanation of the study protocol, purpose and methodology including the difference between the two study groups. Willing participants will sign an informed consent.
2. At the initiation visit, the patient will be randomly assigned to one of the two study groups.
3. Following the random assignment, all participants will complete 3 validated questionnaires. The first questionnaire, validated to a state of acute anxiety, termed STAI:Y-1, The State-Trait Anxiety Inventory. This version, includes 20 items representing anxiety related sensations. Patients will be instructed to scale on a range of 1 to 4, where 1 stands for strongly disagree and 4 for strongly agree, how do each of the items represent the current state of anxiety. The final grade for each questionnaire is obtained through summing all ranks. The scale is reversed for each item phrased in a positive note before summation.

   A higher grade correlates with greater anxiety. Addendum 1. The second questionnaire validated to the evaluation of maternal attachment to the fetus during pregnancy until the week of recruitment to the study. The questionnaire is termed: Maternal Antenatal Attachment Scale-MAAS (female) Addendum 2. The third questionnaire, validated to evaluate the overall pregnancy experience: Revised Prenatal Distress Questionnaire (NUPDQ; Lobel et al., 2008) Addendum 3.

   After completion of the questionnaires, the patients will be instructed on the mode of operation of home ultrasound device (pulsenmore), the frequency and means of communication with the study team. The patient will receive a written manual of operation for the device and will sign a contract obligating to preserve and return the device at the end of the study period.
4. At 20-22 weeks of gestation, the participants will complete again all the three questionnaires. During that visit, the patient will return the device to the present team member.
5. Collected data includes:

   1. Demographic characteristics (age, BMI, smoking, number of pregnancies, number of deliveries, past obstetrical and medical history, use of medication)
   2. Antenatal follow-up
   3. The results of the various questionnaires primary outcome The delta between The State-Trait Anxiety Inventory (STAI:Y-1) score filled at recruitment and at 20-22 weeks of gestation (when patient start fill fetal movements).

Secondary outcomes The delta between The Maternal Antenatal Attachment Scale MAAS and the Distress Questionnaire score filled at recruitment and at 20-22 weeks of gestation.

Number of obstetric ICU referrals Number of admissions for hospitalization during pregnancy

Sample size For the purpose of calculating the sample size, suppose that The State-Trait Anxiety Inventory (STAI: Y-1) at the second trimester for a patient with reccurent pregnancy losses is 40 units with a standard deviation of 5 units based on previous work. 9 to demonstrate a decrease in the score) The State-Trait Anxiety Inventory (STAI: Y-1) in 8 units will need to recruit 50 women (25 per group) with 80 percent power and 0.05 alpha.

Research funding - The authors will not receive any financial support for the research.

The devices are provided as a contribution for the research period by the Pulsenmore Company

Study Duration - 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recurrent pregnancy losses in first trimester
2. Current pregnancy gestational age 12-14 week of gestation
3. Singleton pregnancy

Exclusion Criteria:

1. Female subjects who refuse to participate
2. Female subjects who don't speak Hebrew

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-12-23 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety levels | 10 weeks
  The delta between The State-Trait Anxiety Inventory (STAI:Y-1) score filled at recruitment and at 20-22 weeks of gestation (when patient start fill fetal movements).

CONTACTS AND LOCATIONS:
Overall Officials: Michal Levi, Dr., Principal Investigator — Wolfson Medical Center
Locations (1):
- Departments of Obstetrics & Gynecology, affiliated with Sackler Faculty of Medicine, Tel Aviv University, Holon, Israel

REFERENCES:
- [Background] Macklon NS, Geraedts JP, Fauser BC. Conception to ongoing pregnancy: the 'black box' of early pregnancy loss. Hum Reprod Update. 2002 Jul-Aug;8(4):333-43. doi: 10.1093/humupd/8.4.333. PMID 12206468
- [Background] Practice Committee of the American Society for Reproductive Medicine. Definitions of infertility and recurrent pregnancy loss: a committee opinion. Fertil Steril. 2013 Jan;99(1):63. doi: 10.1016/j.fertnstert.2012.09.023. Epub 2012 Oct 22. PMID 23095139
- [Background] Lee C, Slade P. Miscarriage as a traumatic event: a review of the literature and new implications for intervention. J Psychosom Res. 1996 Mar;40(3):235-44. doi: 10.1016/0022-3999(95)00579-x. PMID 8861119
- [Background] Bergner A, Beyer R, Klapp BF, Rauchfuss M. Pregnancy after early pregnancy loss: a prospective study of anxiety, depressive symptomatology and coping. J Psychosom Obstet Gynaecol. 2008 Jun;29(2):105-13. doi: 10.1080/01674820701687521. PMID 17943588
- [Background] Lee C, Slade P, Lygo V. The influence of psychological debriefing on emotional adaptation in women following early miscarriage: a preliminary study. Br J Med Psychol. 1996 Mar;69(1):47-58. doi: 10.1111/j.2044-8341.1996.tb01849.x. PMID 8829399
- [Background] Woods-Giscombe CL, Lobel M, Crandell JL. The impact of miscarriage and parity on patterns of maternal distress in pregnancy. Res Nurs Health. 2010 Aug;33(4):316-28. doi: 10.1002/nur.20389. PMID 20544819
- [Background] Tsartsara E, Johnson MP. The impact of miscarriage on women's pregnancy-specific anxiety and feelings of prenatal maternal-fetal attachment during the course of a subsequent pregnancy: an exploratory follow-up study. J Psychosom Obstet Gynaecol. 2006 Sep;27(3):173-82. doi: 10.1080/01674820600646198. PMID 17214452
- [Background] Hada K, Kuse E, Nakatsuka M. Women with Recurrent Pregnancy Loss : Their Psychology During Late Pregnancy and the Supportive Behavior of Their Partners. Acta Med Okayama. 2018 Aug;72(4):387-394. doi: 10.18926/AMO/56176. PMID 30140087